CLINICAL TRIAL: NCT05257395
Title: A Phase III Study to Evaluate the Efficacy and Safety of XZP-3287 Combined With Letrozole/Anastrozole Versus Placebo Combined With Letrozole/Anastrozole in Patients With HR Positive and HER2 Negative Recurrent/Metastatic Breast Cancer
Brief Title: A Study of XZP-3287 in Combination With Letrozole/Anastrozole in Patients With Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XZP-3287-3002
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer
Keywords: XZP-3287; HR positive Her2 negative recurrent/metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XZP-3287+ Letrozole/Anastrozole (Experimental)
  Interventions: Drug: XZP-3287+ Letrozole/Anastrozole
- Placebo + Letrozole/Anastrozole (Placebo Comparator)
  Interventions: Drug: Placebo + Letrozole/Anastrozole

INTERVENTIONS:
Drug: XZP-3287+ Letrozole/Anastrozole — XZP-3287 360 mg orally after meals Twice daily of every 28-day cycle; Letrozole tablets 2.5mg orally once daily of every 28-day cycle or Anastrozole tablets 1mg orally once daily of every 28-day cycle
  Arms: XZP-3287+ Letrozole/Anastrozole
Drug: Placebo + Letrozole/Anastrozole — Placebo 360 mg orally after meals Twice daily of every 28-day cycle; Letrozole tablets 2.5mg orally once daily of every 28-day cycle or Anastrozole tablets 1mg orally once daily of every 28-day cycle
  Arms: Placebo + Letrozole/Anastrozole

SUMMARY:
This is a Phase III clinical trial designed to evaluate the efficacy and safety of XZP-3287 in combination with Letrozole/Anastrozole versus placebo in combination with Letrozole/Anastrozole in patients with HR-positive and HER2-negative recurrent/metastatic breast cancer who have not received systemic anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years and ≤75 years old;
2. Patient is in the menopausal state；
3. Histologically or cytologically confirmed locally advanced, recurrent or metastatic breast cancer, which was pathologically confirmed to be HR-positive and HER2-negative;
4. Evidence of locally advanced, recurrent, or metastatic disease that is not amenable to curative surgical resection or radiation therapy and is not clinically amenable to chemotherapy;
5. No prior systemic anticancer therapy for locally advanced, recurrent, or metastatic disease;
6. At least one measurable lesion (based on RECIST v1.1) or only bone metastases;
7. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
8. Adequate organ and marrow function;
9. Patient of childbearing age must undergo a serum pregnancy test within 7 days before randomization, and the result is negative; patient is willing to use a medically approved high-efficiency contraceptive method during the study period and within 6 months after the last study drug treatment;
10. Patient with acute toxic reactions caused by previous anti-tumor treatments or surgical operations were alleviated to grade 0 to 1 (NCI-CTCAE v5.0), or to the level specified by the enrollment criteria;
11. Patient has signed informed consent before any trial related activities.

Exclusion Criteria:

1. Patients with disease recurrence or metastasis at or within 12 months after previous neoadjuvant or adjuvant therapy with endocrine drugs;
2. Patient with visceral crisis or brain metastases, except for patient with stable brain metastases;
3. Patient had clinically significant pleural effusions, ascites effusions, or pericardial effusions in the 4 weeks before enrollment;
4. Patient who received prior treatment with mTOR inhibitors or CDK4/6 inhibitors ;
5. Participation in a prior treatment of major surgery, chemotherapy, radiotherapy, and any anti-tumor treatment within 14 days before enrollment；
6. Patient who participated in other clinical trials within 14 days before enrollment or within 5 half-lives of the trial drug, whichever is longer;
7. Patient used CYP3A4 potent inhibitors or potent inducers within 14 days before enrollment or within 5 half-lives of the drug, whichever is longer;
8. Initiation of bisphosphonates or RANKL inhibitors within 7 days before enrollment, and subjects who have initiated treatment > 7 days before enrollment should not change the method of use;
9. Any other malignant tumor has been diagnosed within 5 years before randomization;
10. Patient is in the active stage of HBV, HCV or co-infected with HBV, HCV, or Patient with positive HIV antibody;
11. Patient with severe infection within 4 weeks before enrollment, or unexplained fever> 38.3℃ during screening/before enrollment;
12. Patient with heart function impaired or clinically significant heart disease within 6 months before enrollment;
13. Cerebrovascular accident occurred within 6 months before enrollment, including history of transient ischemic attack or stroke; pulmonary embolism;
14. Inability to swallow, intestinal obstruction or other factors that affect the taking and absorption of the drug;
15. Patient with a known hypersensitivity to any of the excipients in this study;
16. A prior history of autologous or allogeneic hematopoietic stem cell transplantation;
17. A prior history of psychotropic drug abuse or drug use;
18. Nursing Mothers;
19. The researchers considered that there were some cases that were not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2030-09-05 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed progression free survival (PFS) | Up to approximately 24 months

SECONDARY OUTCOMES:
BICR-assessed progression free survival (PFS) | Up to approximately 24 months
Overall survival (OS) | Up to approximately 5 years
Overall survival rate(OSR) | Up to approximately 5 years
Objective response rate (ORR) | Up to approximately 24 months
Duration of response (DoR) | Up to approximately 24 months
Disease control rate (DCR) | Up to approximately 24 months
Clinical benefit rate (CBR) | Up to approximately 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to approximately 24 months
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | Up to approximately 24 months
Maximum Plasma Concentration [Cmax] | Up to approximately 4 months
Time to Maximum Plasma Concentration [Tmax] | Up to approximately 4 months
Area under the time-concentration Curve [AUC] | Up to approximately 4 months

OTHER OUTCOMES:
Time to Deterioration（TTD） | Up to approximately 24 months
  Time from randomization to the first worsening of the EORTC QLQ-C30 scale score.
EORTC QLQ-C30 scale | Up to approximately 24 months
EORTC QLQ-BR23 scale | Up to approximately 24 months
EQ-5D-5L scale | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhang, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University
Locations (1):
- Harbin Medical University Cancer Hospital, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No
The data supporting the findings of this trial, including source data, cannot be made available openly owing to their proprietary nature and that the BRIGHT-3 study is still ongoing and blinded.